CLINICAL TRIAL: NCT00593151
Title: An Open-Label, 3-Panel, Dose-Escalation Study to Assess the Safety and Tolerability, Pharmacokinetics, and Viral Kinetics of Two Doses of LocteronTM (Poly ActiveTM - Interferon Alpha 2b) Given Every 2 Weeks for 4-12 Weeks in Comparison With PEG-Intron Given Weekly for 4-12 Weeks in Patients With Chronic Hepatitis C
Brief Title: Study of Safety, Tolerability, and Anti-Viral Effect of Locteron Compared to PEG-Intron in Patients With Chronic Hepatitis C
Acronym: PLUS
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Biolex Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S07-200-02-003
Record Dates: First submitted 2008-01-02; First posted 2008-01-14 (Estimated); Last update posted 2012-02-03 (Estimated); Status verified 2012-02

CONDITIONS: Hepatitis C
Keywords: Antimetabolites; Virus Diseases; Anti-Infective Agents; RNA Virus Infections; Digestive System Diseases; Flaviviridae Infections; Antineoplastic Agents; Therapeutic Uses; Antiviral Agents; Molecular Mechanisms of Action; Pharmacologic Actions
MeSH Terms: conditions — Hepatitis C; Virus Diseases; RNA Virus Infections; Digestive System Diseases; Flaviviridae Infections | interventions — locteron; peginterferon alfa-2b

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- A, C, 320 mcg (Experimental): Bi-weekly subcutaneous doses of Locteron (controlled-release interferon alpha 2b) with oral ribavirin.
  Interventions: Other: Locteron (controlled-release interferon alpha 2b)
- B, C, 640 mcg (Experimental): Bi-weekly subcutaneous doses of Locteron (controlled-release interferon alpha 2b) with oral ribavirin.
  Interventions: Other: Locteron (controlled-release interferon alpha 2b)
- A, B, C PEG (Active Comparator): Weekly subcutaneous injections of 1.5 ug/kg PegIntron (12 kDalton pegylated interferon alpha 2b) with oral ribavirin.
  Interventions: Biological: pegylated IFNa2b

INTERVENTIONS:
Other: Locteron (controlled-release interferon alpha 2b) — biological+device, bi-weekly subcutaneous injections for 4-12 weeks, 160 mcg per injection
  Other Names: PolyActive-IFNa2b; BLX-883+PolyActive
  Arms: A, C, 320 mcg; B, C, 640 mcg
Biological: pegylated IFNa2b — biological, weekly subcutaneous injections for 4-12 weeks, 1.5 mcg/kg
  Other Names: PEG-Intron; PEG; 12 kDalton pegylated interferon alpha 2b
  Arms: A, B, C PEG

SUMMARY:
The purposes of the PLUS study were to confirm the safety and tolerability of two doses of LocteronTM (320 ug and 640 ug) dosed over four weeks in patients who had failed prior anti-HCV therapies (Panels A and B), and then to continue to study the safety, tolerability, and preliminary efficacy of the same two doses of LocteronTM (320 ug and 640 ug) in treatment-naïve genotype 1 HCV patients when Locteron dosed over 12 weeks (Panel C). All subjects were also to receive oral daily weight-based ribavirin.

DETAILED DESCRIPTION:
Panels A and B of the PLUS study were designed to assess the safety and tolerability, pharmacokinetics, and viral kinetics over four weeks of two doses of Locteron™ (230 ug and 640 ug) given every two weeks in comparison with PegIntron® given weekly in treatment-experienced subjects with chronic hepatitis C of any genotype who were co-administered weight-based oral ribavirin. The two cohorts of 16 subjects each in Panels A and B consisted of subjects who had failed prior interferon therapy. In Panel A, 8 subjects were randomized to and completed 4 weeks of treatment with 320 μg Locteron™ and 8 subjects were randomized to and completed 4 weeks of treatment with 1.5 ug/kg PegIntron®. In Panel B, 8 subjects were randomized to and completed 4 weeks of treatment with 640 μg Locteron™ and 8 subjects were randomized to and completed 4 weeks of treatment with 1.5 ug/kg PegIntron®. When the results of Panel A and Panel B were known, conduct of Panel C for 12 weeks in treatment-naive patients with chronic genotype-1 HCV was considered unnecessary and cancelled, and an entirely new study was begun instead.

ELIGIBILITY:
Inclusion Criteria:

* Evidence of chronic hepatitis C
* Positive HCV RNA test with a level >= 1 x 104 IU/mL (by RT-PCR)

Exclusion Criteria:

* Decompensated Liver Disease
* Positive test for serum antibodies to the human immunodeficiency virus (HIV), hepatitis A (HAV-IgM), o hepatitis B (HBV- +Hepatitis B surface antigen)
* A history of severe psychiatric disease, including major depression
* A history of immunologically-mediated disease, COPD, severe asthma, severe cardiac disease, active cancer or cancer within last 5 years, seizures within the past 5 years or epilepsy, solid organ or bone marrow transplant, uncontrolled thyroid disease, or clinically significant retinopathy
* Pregnant or lactating females

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2008-01; Primary Completion 2008-12 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
To assess in subjects with chronic hepatitis C the safety and tolerability of Locteron in comparison with PEG-Intron. | 7 months (4 weeks of treatment, 6 months of follow up)

SECONDARY OUTCOMES:
To assess in subjects with chronic hepatitis C receiving a weight-based oral daily dose of ribavirin: • The PK profile of Locteron (IFNa2b) • The preliminary efficacy of Locteron assessed by serial quantitation of HCV RNA levels | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Walker Long, MD, Study Director — Biolex Therapeutics, Inc.
Locations (5):
- United States (5):
  - Henry Ford Hospital, Detroit, Michigan
  - Methodist Dallas Medical Center, Dallas, Texas
  - Alamo Medical Research, San Antonio, Texas
  - Inova Center for Liver Diseases, Annandale, Virginia
  - McGuire DVAMC, McGuire Research Institute, Richmond, Virginia

REFERENCES:
- [Result] Lawitz E, Younossi ZM, Shiffman M, Gordon S, Ghalib R, Long W, Muir A, McHutchison J. Randomized trial comparing systemic and local reactions to controlled-release interferon alpha2b and pegylated-interferon alpha2b in hepatitis C subjects who failed prior treatment. J Hepatology 50:S231 (abstract 628), 2009. (Presented to the 44th Annual Meeting Of The European Association for the Study of the Liver, April 22-26, 2009.)